CLINICAL TRIAL: NCT00288275
Title: A Non-Interventional Prospective Study of the Correlation of the Precision Therapeutics, Inc. Chemoresponse Assay With Progression-Free Survival in Patients With Recurrent Epithelial Ovarian, Peritoneal, or Fallopian Tube Cancer.
Brief Title: Correlation of the Chemoresponse Assay With PFS in Patients With Recurrent Epithelial Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Terminated | Type: Observational
Sponsor: Precision Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PT-301; NCT00301717 (obsolete NCT alias)
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Assay; Chemotherapy; Recurrent; Refractory; Persistent; Chemoresponse; Sensitivity; Precision Therapeutics
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Recurrence; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover tumor cells from the test, pathology slides, and blood samples will be collected and stored to look for potential genetic variations related to drug pathway genes to identify patterns associated with clinical outcome.

SUMMARY:
Chemoresponse assays (lab test) measure the effect that chemotherapy treatment has on a patient's cancer cells in the lab. This test has shown success in a retrospective study in predicting how an individual patient's tumor will respond to a given chemotherapy and how treatment utilizing an agent that the test said that a patient's cells would be sensitive too corresponds to a longer progression free interval. This study will determine the ability of two tests used to predict the success of chemotherapy in recurrent, persistent, or refractory cancer of the ovaries, fallopian tube(s) or peritoneum by measuring how long patients live without progression.

DETAILED DESCRIPTION:
The traditional treatment course for new cases of ovarian, fallopian tube, or peritoneal cancer is cytoreductive surgery followed by chemotherapy with paclitaxel in combination with carboplatin. Unfortunately, despite high initial response rates, the majority of patients recur and subsequent therapy is much less likely to be effective. The use of ineffective chemotherapy can result in unnecessary toxicity and costs, delay of more effective treatment, and the potential for the development of cross-resistance to additional drugs. The ability to individualize therapy by providing the treating physician with ex vivo response information on a panel of drugs should aid in the selection of effective therapy for individual patients, thus resulting in improved outcomes.

Resistance to chemotherapy cannot be predicted by either clinical or histological examination. Historically, the ex vivo sensitivity and resistance of tumor cells has been evaluated as a tool for predicting the clinical response of the patient to therapy. In this study, chemotherapy drugs will be tested using both the Precision Therapeutics' ChemoFx Assay and the Yale Apoptosis Assay. The assay results will be compared to clinical outcomes that will be reported at regular intervals. Blood, tumor pathology slides, and excess tumor cells (if available) will be used to characterize common polymorphisms in drug metabolizing enzymes as well as other molecular markers potentially associated with tumor response.

This is a one-arm validation trial with a goal of approximately 256 evaluable patients recruited from multiple sites. Patients will be drawn from the Yale -New Haven Medical Center and multiple additional sites as needed to meet accrual goals. The patients will be treated with FDA approved drugs and/or drug combinations based on the medical judgment of the treating physician. The study is not randomized and the results of the assay will not be used in the decision process for which agent to select for treatment, but are made available to the treating physician upon further progression.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with persistent, refractory, or recurrent epithelial ovarian, peritoneal, or fallopian tube carcinoma.
* Patient must have documented disease defined by physical exam, clinically significant increases in CA-125 (as defined by protocol), CT, MRI scan, PET, x-ray or ultrasound for whom cytoreduction, excisional biopsy, incisional biopsy, or paracentesis is medically indicated, or in the alternative, have agreed to a core biopsy of the primary site, a secondary metastatic site, or a paracentesis or thoracentesis for fluid collection.
* Patient has disease of one of the following histologic epithelial cell types: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, transitional cell carcinoma, clear cell carcinoma, or adenocarcinoma, not otherwise specified (N.O.S.). Cytologic confirmation of diagnosis is acceptable for patients treated with neoadjuvant therapy who have not had a surgical procedure for a histologic confirmation.
* Patient has only received one or two prior chemotherapy regimens for their ovarian, peritoneal, or fallopian tube carcinoma. Multiple previous regimens of Taxol/Carboplatin will be counted as 1 prior chemotherapy regimen (e.g., A patient who receives first line Taxol/Carboplatin, then recurs, then receives Taxol/Carboplatin will be considered to have had only 1 prior regimen.)
* Patient must have completed prior chemotherapy regimens at least 3 weeks prior to tissue extraction.
* Patient must have an estimated life expectancy of greater than six months, as determined by the investigator.
* Patient requires chemotherapy and the investigator plans to administer one of the regimens of interest as deemed by her physician.
* Patient must be a female and at least 18 years of age. Ovarian cancer is a disease that occurs only in women and is exceedingly rare in females under the age of 18.
* Patient must have an ECOG Performance Status of 0, 1, or 2.
* Tumor tissue or ascitic fluid must be available for the assays. Ascites or Pleural alone may be collected and submitted as the sample tissue, but the patient must also have measurable disease as demonstrated by a CA-125 level 2X ULN or measurable lesions on imaging to be eligible.
* Patient must have signed an approved consent form.

Exclusion Criteria:

* Patient has ovarian stromal, mixed mullerian, or germ cell tumors
* Patient has borderline carcinoma (uncertain malignant potential)
* Pregnant or lactating patients
* Patients of childbearing potential not employing adequate contraception.
* Patients who are at risk of failure of compliance to the visit schedules and procedures.
* The investigator plans to use an assay to select the chemotherapy drug regimen. The investigator may submit the patient's tissue for testing with other assays, but may not use the results of those assays to select the chemotherapy regimen for the patient for this trial.
* Patients with synchronous primary endometrial cancer or a past history of primary endometrial cancer are excluded unless all of the following conditions are met: Stage not greater than I-B, Less than 3mm invasion without vascular or lymphatic invasion, NO poorly differentiated subtype, including papillary serous, clear cell, or othe FIGO Grade 3 lesion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 500 patients will be enrolled at 20-30 US sites. Patients have been diagnosed with persistent, refractory, or recurrent epithelial ovarian, peritoneal, or fallopian tube cancer.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2004-07; Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 1. Every Treatment Cycle 2. Every 3 months for the first 2 years post treatment 3. Every 6 months for the next 3 years post treatment 4. Annually thereafter.

SECONDARY OUTCOMES:
Tumor Response | 1. Every treatment cycle 2. Every 3 months for the first 2 years post treatment 3. Every 6 months for the next 3 years post treatment 4. Annually thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Rutherford, MD, Principal Investigator — Yale University; Hong Ma, MD, Study Director — Precision Therapeutics, Inc.
Locations (36):
- United States (36):
  - University of California, Irvine, California
  - Kaiser Permanente, Los Angeles, California
  - Yale University Medical Center, New Haven, Connecticut
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - St. Vincents Medical Center, Jacksonville, Florida
  - The Florida Hospital, Orlando, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - Southeastern Gynecologic Oncology Riverdale, Riverdale, Georgia
  - Northwestern University/Prentice Women's Hospital, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - The Cooper Health System, Camden, New Jersey
  - Saint Barnabas Medical Center, West Orange, New Jersey
  - Schwartz Gynecologic Oncology, PLLC, Brightwaters, New York
  - University of Cincinnati Medical Center Barrett Cancer Center, Cincinnati, Ohio
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Health System, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Cancer Center at Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Mainline Health System, Wynnwood, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - ACORN - The West Clinic, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin, Madison, Madison, Wisconsin

REFERENCES:
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Background] Ness RB, Wisniewski SR, Eng H, Christopherson W. Cell viability assay for drug testing in ovarian cancer: in vitro kill versus clinical response. Anticancer Res. 2002 Mar-Apr;22(2B):1145-9. PMID 12168915
- [Background] O'Meara AT, Sevin BU. Predictive value of the ATP chemosensitivity assay in epithelial ovarian cancer. Gynecol Oncol. 2001 Nov;83(2):334-42. doi: 10.1006/gyno.2001.6395. PMID 11606094
- [Background] McLeod HL, King CR, Marsh S. Application of pharmacogenomics in the individualization of chemotherapy for gastrointestinal malignancies. Clin Colorectal Cancer. 2004 Jun;4 Suppl 1:S43-7. doi: 10.3816/ccc.2004.s.007. PMID 15212705
- [Background] Kaplan EL, Meier P. Nonparametric estimation of incomplete observations. JASA 1958;43:457-481.
- [Background] Journal of Clinical Oncology, 2004 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 22, No 14S (July 15 Supplement), 2004: 5074.